CLINICAL TRIAL: NCT03224676
Title: Study to Assess the Quality of Sleep and Perceived Sleep Distractors Among the Adult Patients Admitted in Selected Hospital
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, priti sirohi, Student, M.sc. Nursing, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: IEC/P.N786
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Quality of Sleep
Keywords: Quality of sleep; Perceived sleep distractors; Adult patients
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study was to assess the quality of sleep among adult patients, to explore the perceived sleep distractors among adult patients, to determine the relationship between quality of sleep and perceived sleep distractors score among adult patients.

and to determine the association of quality of sleep and perceived sleep distractors score among adult patients with selected variables.

DETAILED DESCRIPTION:
A total of 150 adult patients were selected from surgical, orthopedic and medical wards to participate in the study 50 patients from each ward. All the adult patients were selected using convenience sampling technique. Self-introduction and establishing rapport with the subjects was done. Purpose of the study was explained to the subjects, the confidentially of their responses was assured, and informed consent was taken prior to the study. The data was collected by Modified Pittsburgh Sleep Quality Index and Structured Perceived Sleep Distractors Performa.

ELIGIBILITY:
Inclusion Criteria:

The study includes adult patients who were:

* between age group of 18-65 years
* hospitalized minimum for 7 days.
* willing to participate in the study.
* present at the time of data collection.

Exclusion Criteria:Adult patients who were not:

* alert and oriented.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of sleep | 20-25 min.
  It comprised of total 7 components. Each item is rated as 0, 1, 2, 3. The maximum possible score was 21 and minimum possible score was zero on the Modified Pittsburgh sleep Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Sirohi, Msc.Nursing, Principal Investigator — Maharishi Markandeshwar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levenson JC, Shensa A, Sidani JE, Colditz JB, Primack BA. The association between social media use and sleep disturbance among young adults. Prev Med. 2016 Apr;85:36-41. doi: 10.1016/j.ypmed.2016.01.001. Epub 2016 Jan 11. PMID 26791323
- [Background] van Leeuwen WM, Lehto M, Karisola P, Lindholm H, Luukkonen R, Sallinen M, Harma M, Porkka-Heiskanen T, Alenius H. Sleep restriction increases the risk of developing cardiovascular diseases by augmenting proinflammatory responses through IL-17 and CRP. PLoS One. 2009;4(2):e4589. doi: 10.1371/journal.pone.0004589. Epub 2009 Feb 25. PMID 19240794
- [Background] Shim J, Kang SW. Behavioral Factors Related to Sleep Quality and Duration in Adults. J Lifestyle Med. 2017 Jan;7(1):18-26. doi: 10.15280/jlm.2017.7.1.18. Epub 2017 Jan 31. PMID 28261557